CLINICAL TRIAL: NCT03563482
Title: Correlazione Dell'Imaging Metabolico Con l'Espressione Dei Marcatori Immunitari Nei Pazienti Con NSCLC Candidati All'Immunoterapia.
Brief Title: Correlation of Metabolic Imaging With Immune Markers in NSCLC Candidate to Immunotherapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1670
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Positron-Emission Tomography; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Positron-Emission Tomography; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Biopsy and PET scan
  Interventions: Diagnostic Test: PET scan

INTERVENTIONS:
Diagnostic Test: PET scan — Tumor biopsy at baseline; PET scan performed after 8 weeks of treatment
  Other Names: Biopsy

SUMMARY:
The purpose of the present study is to prospectively investigate the correlation between the metabolic parameters on FDG-PET before and during immunotherapy treatment with the immune infiltrate and other tissue or circulating markers in a NSCLC patients candidate to immunotherapy.

DETAILED DESCRIPTION:
This is an interventional prospective study without medication lasting 36 months, including an estimated period of 18 months for the enrolment and max 18 months of follow-up. All consecutive patients affected by NSCLC and referred for immunotherapy with the anti-PD-1 agent nivolumab, or other checkpoint inhibitors that may become available in the future, will be prospectively enrolled. The study cohort will consist of 40 patients.

All patients will undergo the following steps: 1) selection based on eligibility criteria and informed consent; 2) baseline examinations (ceCT and 18F-FDG PET/CT); 3) tumor biopsy and blood sampling; 4) Immunotherapy with check-point inhibitors; 5) response evaluation after 8 weeks of treatment (ceCT and 18F-FDG PET/CT) and second blood sampling; 6) follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients with pathological diagnosis of NSCLC eligible for immunotherapy;
* obtained informed consent.

Exclusion Criteria:

* age <18 years;
* pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlate the tumor expression of immune markers with the metabolic characteristics on FDG-PET in patients with NSCLC candidates to immunotherapy. | Baseline
  Standardized uptake value

SECONDARY OUTCOMES:
Tumor expression of immune markers with the metabolic characteristics on FDG-PET in patients with NSCLC candidates to immunotherapy. | Before treatment
  Metabolic tumor burden
Correlate immune markers with the metabolic characteristics on FDG-PET in patients with NSCLC candidates to immunotherapy. | Baseline
  Tumor infiltrate
Evaluate the variation of metabolic parameters on FDG-PET in patients with NSCLC before and 8 weeks after the first administration of immunotherapy. | After 8 weeks of treatment
  Standardized uptake value
Quantify the variation of metabolic parameters on FDG-PET in patients with NSCLC before and 8 weeks after the first administration of immunotherapy. | After 8 weeks of treatment
  Metabolic tumor burden
Evaluate other tissue or circulating markers in patients with NSCLC before and 8 weeks after the first administration of immunotherapy. | Baseline
  Tissue and blood samples
Evaluate other tissue or circulating markers in patients with NSCLC before and 8 weeks after the first administration of immunotherapy. | 8 weeks after treatment
  Tissue and blood samples

OTHER OUTCOMES:
Correlate all defined parameters with response to treatment and outcome | 18 months of follow up
  Response assessment and disease outcome

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castello A, Grizzi F, Toschi L, Rossi S, Rahal D, Marchesi F, Russo C, Finocchiaro G, Lopci E. Tumor heterogeneity, hypoxia, and immune markers in surgically resected non-small-cell lung cancer. Nucl Med Commun. 2018 Jul;39(7):636-644. doi: 10.1097/MNM.0000000000000832. PMID 29608508
- [Background] Grizzi F, Castello A, Lopci E. Is it time to change our vision of tumor metabolism prior to immunotherapy? Eur J Nucl Med Mol Imaging. 2018 Jun;45(6):1072-1075. doi: 10.1007/s00259-018-3988-1. Epub 2018 Mar 12. No abstract available. PMID 29532102
- [Background] Rossi S, Toschi L, Castello A, Grizzi F, Mansi L, Lopci E. Clinical characteristics of patient selection and imaging predictors of outcome in solid tumors treated with checkpoint-inhibitors. Eur J Nucl Med Mol Imaging. 2017 Dec;44(13):2310-2325. doi: 10.1007/s00259-017-3802-5. Epub 2017 Aug 16. PMID 28815334
- [Background] Lopci E, Toschi L, Grizzi F, Rahal D, Olivari L, Castino GF, Marchetti S, Cortese N, Qehajaj D, Pistillo D, Alloisio M, Roncalli M, Allavena P, Santoro A, Marchesi F, Chiti A. Correlation of metabolic information on FDG-PET with tissue expression of immune markers in patients with non-small cell lung cancer (NSCLC) who are candidates for upfront surgery. Eur J Nucl Med Mol Imaging. 2016 Oct;43(11):1954-61. doi: 10.1007/s00259-016-3425-2. Epub 2016 Jun 1. PMID 27251642
- [Background] Castello A, Toschi L, Rossi S, Mazziotti E, Lopci E. The immune-metabolic-prognostic index and clinical outcomes in patients with non-small cell lung carcinoma under checkpoint inhibitors. J Cancer Res Clin Oncol. 2020 May;146(5):1235-1243. doi: 10.1007/s00432-020-03150-9. Epub 2020 Feb 11. PMID 32048008
- [Background] Rossi S, Castello A, Toschi L, Lopci E. Immunotherapy in non-small-cell lung cancer: potential predictors of response and new strategies to assess activity. Immunotherapy. 2018 Jul;10(9):797-805. doi: 10.2217/imt-2017-0187. PMID 30008262
- [Background] Castello A, Lopci E. Response assessment of bone metastatic disease: seeing the forest for the trees RECIST, PERCIST, iRECIST, and PCWG-2. Q J Nucl Med Mol Imaging. 2019 Jun;63(2):150-158. doi: 10.23736/S1824-4785.19.03193-5. Epub 2019 Jul 8. PMID 31286751
- [Background] Castello A, Rossi S, Mazziotti E, Toschi L, Lopci E. Hyperprogressive Disease in Patients with Non-Small Cell Lung Cancer Treated with Checkpoint Inhibitors: The Role of 18F-FDG PET/CT. J Nucl Med. 2020 Jun;61(6):821-826. doi: 10.2967/jnumed.119.237768. Epub 2019 Dec 20. PMID 31862803
- [Background] Monterisi S, Castello A, Toschi L, Federico D, Rossi S, Veronesi G, Lopci E. Preliminary data on circulating tumor cells in metastatic NSCLC patients candidate to immunotherapy. Am J Nucl Med Mol Imaging. 2019 Dec 15;9(6):282-295. eCollection 2019. PMID 31976158
- [Background] Castello A, Carbone FG, Rossi S, Monterisi S, Federico D, Toschi L, Lopci E. Circulating Tumor Cells and Metabolic Parameters in NSCLC Patients Treated with Checkpoint Inhibitors. Cancers (Basel). 2020 Feb 19;12(2):487. doi: 10.3390/cancers12020487. PMID 32092983
- [Background] Castello A, Lopci E. Update on tumor metabolism and patterns of response to immunotherapy. Q J Nucl Med Mol Imaging. 2020 Jun;64(2):175-185. doi: 10.23736/S1824-4785.20.03251-3. Epub 2020 Feb 27. PMID 32107904
- [Background] Castello A, Rossi S, Toschi L, Mansi L, Lopci E. Soluble PD-L1 in NSCLC Patients Treated with Checkpoint Inhibitors and Its Correlation with Metabolic Parameters. Cancers (Basel). 2020 May 27;12(6):1373. doi: 10.3390/cancers12061373. PMID 32471030
- [Background] Castello A, Rossi S, Toschi L, Lopci E. Comparison of Metabolic and Morphological Response Criteria for Early Prediction of Response and Survival in NSCLC Patients Treated With Anti-PD-1/PD-L1. Front Oncol. 2020 Jul 31;10:1090. doi: 10.3389/fonc.2020.01090. eCollection 2020. PMID 32850315
- [Background] Castello A, Lopci E. Reply: Diagnosis of Hyperprogressive Disease in Patients Treated with Checkpoint Inhibitors Using 18F-FDG PET/CT. J Nucl Med. 2020 Sep;61(9):1405. doi: 10.2967/jnumed.120.243444. Epub 2020 Mar 13. No abstract available. PMID 32169909
- [Background] Lopci E, Haanen JB. Cancer management in the era of immunotherapy: much more than meets the eye. Q J Nucl Med Mol Imaging. 2020 Jun;64(2):141-142. doi: 10.23736/S1824-4785.20.03252-5. Epub 2020 Feb 27. No abstract available. PMID 32107905
- [Background] Aide N, De Pontdeville M, Lopci E. Evaluating response to immunotherapy with 18F-FDG PET/CT: where do we stand? Eur J Nucl Med Mol Imaging. 2020 May;47(5):1019-1021. doi: 10.1007/s00259-020-04702-4. No abstract available. PMID 31996974
- [Background] Aide N, Hicks RJ, Le Tourneau C, Lheureux S, Fanti S, Lopci E. FDG PET/CT for assessing tumour response to immunotherapy : Report on the EANM symposium on immune modulation and recent review of the literature. Eur J Nucl Med Mol Imaging. 2019 Jan;46(1):238-250. doi: 10.1007/s00259-018-4171-4. Epub 2018 Oct 5. PMID 30291373